CLINICAL TRIAL: NCT05598489
Title: Development of Novel Fecal Microbial Biomarkers for Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: National Taiwan University (Other); Hanoi Medical University (Other); Mahidol University (Other); Indonesia University (Other); National University of Malaysia (Other); Kiang Wu Hospital (Other); National Academy of Medical Sciences, Nepal (Other Government); Duke-NUS Graduate Medical School (Other); National University Hospital, Singapore (Other); Heidelberg University (Other); University of Chicago (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: IBDFMB
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease; Microbiome
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Subjects will collect fresh stool in a stool container. Stool DNA will be extracted and stored until used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and Ulcerative colitis (UC), is a chronic idiopathic inflammatory condition of the intestine. Endoscopy has been used to monitor the disease, but it is time-consuming, costly, invasive, and associated with certain risks of morbidity. Many patients are reluctant to undergo repeated endoscopic examinations, particularly when their disease is quiescent. Acute phase reactants have been used to monitor disease including C-reactive protein and stool leucocyte markers including fecal calprotectin, but their sensitivity and specificity in correlating to intestinal inflammation activity are low. Clinical challenge of patient heterogeneity in disease phenotype and response to therapy has compounded discovery of disease-related biomarkers. In IBD, altered fecal microbiota signatures have been consistently reported which included a reduction in biodiversity with lower proportions of Firmicutes and increases in Proteobacteria and Bacteroidetes phylum members. Moreover, overall bacterial diversity is consistently decreased in IBD patients compared to controls. Even though a number of fecal biomarkers have been evaluated for their utility for disease diagnosis in IBD, to date none has been accurate enough for clinical application. Therefore, identification and validation of a non-invasive biomarker which can be easily applied in disease diagnosis and prognosis is warranted to provide an earlier opportunity to intervene. In this study, it aims to develop a metagenomics-based model using fecal microbial biomarkers for differentiating IBD patients from healthy controls, and then validate these fecal microbial biomarkers in different populations.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and Ulcerative colitis (UC), is a chronic idiopathic inflammatory condition of the intestine, which results in diarrhea, rectal bleeding, urgency, weight loss and abdominal pain. The natural course of IBD is characterized by activity outbreaks and periods of remission.

Endoscopy has been used to monitor the disease, but it is time-consuming, costly, invasive, and associated with certain risks of morbidity. Many patients are reluctant to undergo repeated endoscopic examinations, particularly when their disease is quiescent. Acute phase reactants have been used to monitor disease including C-reactive protein and stool leucocyte markers including fecal calprotectin, but their sensitivity and specificity in correlating to intestinal inflammation activity are low. Clinical challenge of patient heterogeneity in disease phenotype and response to therapy has compounded discovery of disease-related biomarkers. In IBD, altered fecal microbiota signatures have been consistently reported which included a reduction in biodiversity with lower proportions of Firmicutes and increases in Proteobacteria and Bacteroidetes phylum members. Moreover, overall bacterial diversity is consistently decreased in IBD patients compared to controls. Even though a number of fecal biomarkers have been evaluated for their utility for disease diagnosis in IBD, to date none has been accurate enough for clinical application. Therefore, identification and validation of a non-invasive biomarker which can be easily applied in disease diagnosis and prognosis is warranted to provide an earlier opportunity to intervene.

In this study, it aims to develop a metagenomics-based model using fecal microbial biomarkers for differentiating IBD patients from healthy controls, and then validate these fecal microbial biomarkers in different populations.

This is a cross-sectional multi-centre study. Two groups of subjects, IBD patients (cases) and healthy subjects (controls), will be recruited from each centre. Each center will provide fecal samples from 80-100 Crohn's disease, 80-100 ulcerative colitis, and 80-100 controls. We will collect clinical data and stool sample from each subject. Fecal microbiota composition will be compared between cases and controls. The abundance of bacterial biomarkers will be assessed, and the efficacy of a diagnostic model will be validated.

ELIGIBILITY:
Cases (Crohn's disease or Ulcerative colitis)

Inclusion Criteria:

* Aged ≥18 years old
* Confirmed diagnosis of Crohn's disease or Ulcerative colitis defined by endoscopy, radiology, and histology
* Competent to provide informed consent

Exclusion Criteria:

* Use of antibiotics in the last 1 month
* Known current sepsis (excluding uncomplicated infections such as influenza)
* Known history of severe organ failure (including decompensated cirrhosis, malignant disease, kidney failure, epilepsy, active serious infection, acquired immunodeficiency syndrome)
* Major bowel surgery in the last 6 months (excluding colonoscopy/ procedure related to perianal disease)
* Presence of an ileostomy / stoma
* Current pregnancy

Controls Inclusion Criteria

* Aged ≥18 years old
* No known medical history including inflammatory bowel disease, irritable bowel syndrome or GI malignancy
* Competent to provide informed consent

Exclusion Criteria

* Use of antibiotics in the last 1 month
* Known current sepsis (excluding uncomplicated infections such as influenza)
* Known history of severe organ failure (including decompensated cirrhosis, malignant disease, kidney failure, epilepsy, active serious infection, acquired immunodeficiency syndrome)
* Bowel surgery in the last 6 months (excluding colonoscopy/ procedure related to perianal disease)
* Presence of an ileos

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases (Crohn's disease or Ulcerative colitis) and healthy controls
Sampling Method: Probability Sample
Enrollment: 3300 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Fecal microbial biomarkers for IBD | 1 year
  To identify and develop fecal microbial biomarkers for IBD, and validate fecal microbial biomarkers in different populations

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong